CLINICAL TRIAL: NCT05059964
Title: Comparison of Circuit Training and Aerobic Exercise on Cardiopulmonary Fitness Among Sedentary Elderly Population
Brief Title: Circuit Training and Aerobic Exercise Among Sedentary Elderly Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REC/01086 Ataur Rahman
Record Dates: First submitted 2021-09-18; First posted 2021-09-28 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Sedentary Behavior; Old Age; Debility
Keywords: Aerobic Exercise; Circuit Training
MeSH Terms: conditions — Sedentary Behavior; Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Circuit Training program (Experimental): circuit training for 4 weeks
  Interventions: Other: Circuit Training program
- Continuous aerobic exercise Group (Active Comparator): aerobic exercise for 4 weeks
  Interventions: Other: Continuous aerobic exercise Group

INTERVENTIONS:
Other: Circuit Training program — The 4 weeks Circuit Training program, it will be of 3 times per week. Each CT workout includes 6 stations per circuit Training. Before the training period, all participants underwent an exercise familiarization session to ensure proper execution of technique.
  The 6 stations will be included as 40 lb. carry for 100 ft., 3-min stair climb, 45 s plank pose, 20 lb. carry with a fast walk for 100 ft., right and left single leg stands for as long as balance was maintained, and a 15 lb. carry up and down 30 stairs
  Arms: Circuit Training program
Other: Continuous aerobic exercise Group — Continuous aerobic exercise Frequency 3 time per week Intensity 50% of Heart rate reserve Type continuous aerobic exercise Time 40 minutes
  Arms: Continuous aerobic exercise Group

SUMMARY:
To compare the effects of Circuit training and aerobic exercise on cardiopulmonary fitness among Sedentary elderly population

ELIGIBILITY:
Inclusion Criteria:

* Participants meeting the below criteria, shall be recruited in the study.
* Sedentary elderly people (Can perform 6 MWT without complication)
* Sedentary elderly population
* No regular exercise or gym activity since last 6 months

Exclusion Criteria:

* Already trained (any gym activity or regular exercise)
* Diagnosed cardiopulmonary disease
* Diabetes
* Any neurological complication

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
6 min walk test: Distance (meters) | 4th Week
  Changes from the baseline, 6 min walk test (6 MWT) was used to measure Functional capacity. It is a sub maximal exercise test which can aid in assessing functional capacity of patients with cardiopulmonary diseases, in this test we find out the maximum distance in meters which an individual covers in 6 min without any support.
Step test | 4th Week
  The Step Test is designed to measure a person's aerobic fitness. Participants step up and down, on and off an aerobics- type step for THREE minutes to increase heart rate and to evaluate the heart's recovery rate during the minute immediately following the step test exercise. Changes from the baseline to 4th week.
  for Age 56-65 heart rate recovery rate in beats per minute fit score: Excellent< 89, Above Average 90-100, Average 101-111, Below Average 112-122, Poor > 123
Forced Expiratory Volume in 1 second (FEV1) | 4th Week
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze Forced Expiratory Volume in 1 second FEV1 in Liters
Forced vital Capacity (FVC) | 4th week
  Changes From the Baseline, the digital spirometer is used in clinical setting to analyze Forced vital Capacity in Liters
Peak Expiratory Flow (PEF) | 4th week
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze peak expiratory flow PEF in Liter/second.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Iqbal Tariq, MSCPPT, Principal Investigator — Riphah International University
Locations (1):
- District Headquarter Hospital - Upper Dir, Dīr, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No